CLINICAL TRIAL: NCT01282593
Title: Potential Role of CD9 and Implication of Motility Process in Pathogenesis of TEL/ALM1-positive ALL Relapses (LAL TEL/ALM1 and CD9).
Acronym: LAL TEL/ALM1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Collaborators: Ligue contre le cancer, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: LOC/10-05; 2010-A00622-37 (Registry Identifier: ID RCB); B100651-40 (Registry Identifier: AFSSAPS reference)
Record Dates: First submitted 2011-01-24; First posted 2011-01-25 (Estimated); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Acute Lymphoblastic Leukemia (ALL)
Keywords: TEL/ALM1_positive ALL relapses
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CD9 expression level (Other): Impact of CD9 expression level on motility assays
  Interventions: Other: Impact of CD9 expression level on motility assays; Other: Post-transcriptional regulation of CD9

INTERVENTIONS:
Other: Impact of CD9 expression level on motility assays — 1) Assess of the impact of CD9 expression level on motility assays (migration and adhesion) We have initiated motility assays (fibronectin adhesion experiments and CXCL12 chemoattracted migration tests with modified Boyden chamber technique) using the CD9 positive TEL/AML1-positive cell line REH and the CD9 negative cell line RAJI (wild or transfected with CD9 cDNA). Data will be analyzed in combination with blocking antibodies and chemical antagonist according to the level of CD9 (transcript and protein) and of CXCR4. Protein quantifications will be performed by flow cytometry and Western Blot. Interactions will be explored by confocal microscopy and biological pathways by immunoblot.
  Adhesion results will be validated on patient samples of B-ALL.
  Other Names: Not Apllicable
Other: Post-transcriptional regulation of CD9 — 2) Post-transcriptional regulation of CD9 in TEL/AML1-positive ALL To identify miRNAs that are potentially deregulated in TEL/AML1-positive acute lymphoblastic leukaemia and especially to screen for CD9 -targeted miRNAs, we will use a TaqMan ®MicroRNA Arrays approach allowing the simultaneous measurement of about 760 human miRNA.
  Small RNA will be extracted from bone marrow samples of twenty childhood B-ALL to screen miRNAs which are differentially expressed between CD9-positive and CD9-negative ALL and further compared with miRNAs which were predicted to target CD9 in databases. Validation of the selection will be performed by single Q-PCR for selected miRNAs using a novel cohort of ten bone marrow samples.
  Other Names: Not Apllicable

SUMMARY:
Down regulation of CD9 in TEL/AML1-positive ALL is addressed in motility assays to explore its role in B-ALL pathogenesis and its potential implication in relapses (and prognosis).

DETAILED DESCRIPTION:
1. Assess of the impact of CD9 expression level on motility assays (migration and adhesion) We have initiated motility assays (fibronectin adhesion experiments and CXCL12 chemoattracted migration tests with modified Boyden chamber technique) using the CD9 positive TEL/AML1-positive cell line REH and the CD9 negative cell line RAJI (wild or transfected with CD9 cDNA). Data will be analyzed in combination with blocking antibodies and chemical antagonist according to the level of CD9 (transcript and protein) and of CXCR4. Protein quantifications will be performed by flow cytometry and Western Blot. Interactions will be explored by confocal microscopy and biological pathways by immunoblot.

   Adhesion results will be validated on patient samples of B-ALL.
2. Post-transcriptional regulation of CD9 in TEL/AML1-positive ALL To identify miRNAs that are potentially deregulated in TEL/AML1-positive acute lymphoblastic leukaemia and especially to screen for CD9 -targeted miRNAs, we will use a TaqMan ®MicroRNA Arrays approach allowing the simultaneous measurement of about 760 human miRNA.

Small RNA will be extracted from bone marrow samples of twenty childhood B-ALL to screen miRNAs which are differentially expressed between CD9-positive and CD9-negative ALL and further compared with miRNAs which were predicted to target CD9 in databases. Validation of the selection will be performed by single Q-PCR for selected miRNAs using a novel cohort of ten bone marrow samples. Transfection assays and luciferase assays will be further realized to confirm that the differential miRNAs really target and affect CD9 expression .

ELIGIBILITY:
Inclusion Criteria:

* patients > 1 year and ≤18 years
* with B-ALL diagnosis
* registered in Rennes for treatment
* written informed consent signed by all patients or their parents or legal guardian

Exclusion Criteria:

* Refusal to participate
* Inherited cytogenetic abnormalities

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 51 (Actual)
Dates: Start 2010-11 (Actual); Primary Completion 2018-10-11 (Actual); Study Completion 2018-10-11 (Actual)

PRIMARY OUTCOMES:
The potential discriminating state of CD9. - To determine the functional impact of CD9 on motility assays in TEL/AML1-positive blasts - To explore the regulation of the expression of the CD9 transcript inTEL/AML1-positive blasts | 3 years
  Due to the importance of the motility process in malignant cells and the role of CD9 in cell motility regulation, we considered the potential discriminating state of CD9.
  * To determine the functional impact of CD9 on motility assays in TEL/AML1-positive blasts
  * To explore the regulation of the expression of the CD9 transcript inTEL/AML1-positive blasts

SECONDARY OUTCOMES:
- Migratory potential of blasts according to CD9 expression | 3 years
  - Migratory potential of blasts according to CD9 expression
- Adhesion properties of blasts according to CD9 expression | 3 years
  - Adhesion properties of blasts according to CD9 expression
- Level of miRNA, that could affect CD9 transcript levels inTEL/AML1-positive blasts versus TEL/AML1-negative ones | 3 years
  - Level of miRNA, that could affect CD9 transcript levels inTEL/AML1-positive blasts versus TEL/AML1-negative ones

CONTACTS AND LOCATIONS:
Locations (1):
- Rennes University Hospital, Rennes, France

REFERENCES:
- [Result] Debaize L, Jakobczyk H, Avner S, Gaudichon J, Rio AG, Serandour AA, Dorsheimer L, Chalmel F, Carroll JS, Zornig M, Rieger MA, Delalande O, Salbert G, Galibert MD, Gandemer V, Troadec MB. Interplay between transcription regulators RUNX1 and FUBP1 activates an enhancer of the oncogene c-KIT and amplifies cell proliferation. Nucleic Acids Res. 2018 Nov 30;46(21):11214-11228. doi: 10.1093/nar/gky756. PMID 30500954
- [Result] Arnaud MP, Vallee A, Robert G, Bonneau J, Leroy C, Varin-Blank N, Rio AG, Troadec MB, Galibert MD, Gandemer V. CD9, a key actor in the dissemination of lymphoblastic leukemia, modulating CXCR4-mediated migration via RAC1 signaling. Blood. 2015 Oct 8;126(15):1802-12. doi: 10.1182/blood-2015-02-628560. Epub 2015 Aug 28. PMID 26320102
- [Result] Gaudichon J, Jakobczyk H, Debaize L, Cousin E, Galibert MD, Troadec MB, Gandemer V. Mechanisms of extramedullary relapse in acute lymphoblastic leukemia: Reconciling biological concepts and clinical issues. Blood Rev. 2019 Jul;36:40-56. doi: 10.1016/j.blre.2019.04.003. Epub 2019 Apr 17. PMID 31010660
- [Result] Rouger-Gaudichon J, Cousin E, Jakobczyk H, Debaize L, Rio AG, Forestier A, Arnaud MP, Villacreces A, Praloran V, Jacamo R, Galibert MD, Troadec MB, Gandemer V. Hypoxia regulates CD9 expression and dissemination of B lymphoblasts. Leuk Res. 2022 Dec;123:106964. doi: 10.1016/j.leukres.2022.106964. Epub 2022 Sep 28. PMID 36335655
- [Result] Debaize L, Jakobczyk H, Rio AG, Gandemer V, Troadec MB. Optimization of proximity ligation assay (PLA) for detection of protein interactions and fusion proteins in non-adherent cells: application to pre-B lymphocytes. Mol Cytogenet. 2017 Jul 20;10:27. doi: 10.1186/s13039-017-0328-2. eCollection 2017. PMID 28736577
- [Result] Jakobczyk H, Debaize L, Soubise B, Avner S, Rouger-Gaudichon J, Commet S, Jiang Y, Serandour AA, Rio AG, Carroll JS, Wichmann C, Lie-A-Ling M, Lacaud G, Corcos L, Salbert G, Galibert MD, Gandemer V, Troadec MB. Reduction of RUNX1 transcription factor activity by a CBFA2T3-mimicking peptide: application to B cell precursor acute lymphoblastic leukemia. J Hematol Oncol. 2021 Mar 20;14(1):47. doi: 10.1186/s13045-021-01051-z. PMID 33743795